CLINICAL TRIAL: NCT00545532
Title: A Double-Blind, Randomized, Stratified Multi-Center Trial Evaluating Conventional and Double Dose Oseltamivir in the Treatment of Immunocompromised Patients With Influenza
Brief Title: A Study of Oseltamivir (Tamiflu) for Treatment of Influenza in Immunocompromised Participants.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NV20234; 2006-002468-24 (EudraCT Number)
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Conventional dose (Experimental): Immunocompromised participants will receive oseltamivir syrup at a dose ranging from 30 to 75 mg based on body weight, twice daily for children (1 to 12 years old) and oseltamivir capsules 75 mg twice daily for adults/adolescents greater than or equal to (>/=) 13 years old or placebo-matched to oseltamivir twice daily over 10 days.
  Interventions: Drug: oseltamivir; Other: placebo
- Double dose (Experimental): Immunocompromised participants will receive oseltamivir syrup at a dose ranging from 60 to 150 mg based on body weight, twice daily for children (1 to 12 years old) and oseltamivir capsules 150 mg twice daily for adults/adolescents (>/=13 years old) or placebo matched to oseltamivir twice daily over 10 days.
  Interventions: Drug: oseltamivir; Other: placebo

INTERVENTIONS:
Drug: oseltamivir — Dose ranging between 30 to 150 mg orally administered as syrup or capsules (depending on participant's age and weight) po twice daily for 10 days
  Other Names: Tamiflu
Other: placebo — Placebo matched to oseltamivir po twice daily for 10 days

SUMMARY:
This 2-arm study will investigate the safety and tolerability of oseltamivir for the treatment of influenza in immunocompromised participants and characterize the effects of oseltamivir in immunocompromised participants on the development of resistant influenza virus. Eligible immunocompromised participants with laboratory-confirmed influenza will be randomized to receive either conventional dose (30 milligrams [mg] to 75 mg twice daily orally [po], depending on age and weight) or double dose (60 mg-150 mg twice daily po depending on age and weight) olseltamivir for 10 days. Nasal and throat swabs will be taken, and safety evaluations made, at intervals during the study. The anticipated time on study medication is 10 days and the anticipated time on study is 40 days.

ELIGIBILITY:
Inclusion Criteria:

* Rapid diagnostic test, PCR, or viral culture positive for influenza in the 96 hours prior to first dose
* Immunocompromised participants with primary or secondary immunodeficiency
* Symptoms suggestive of influenza-like illness
* Use of an effective contraceptive, as specified by protocol; women of childbearing potential cannot be pregnant or breastfeeding

Exclusion Criteria:

* Influenza vaccination with live attenuated vaccine in the 2 weeks prior to randomization
* Antiviral treatment for influenza in 2 weeks prior to randomization
* Severe hepatic impairment
* Any current renal replacement therapy
* Any gastrointestinal disorders which may interfere with the absorption of oseltamivir
* Participation in a study with an investigational drug from 4 weeks prior to study start until study end

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2008-02-04 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (208):
- United States (60):
  - Uni of Alabama At Birmingham; Division of Nephrology, Birmingham, Alabama
  - University of Alabama at Birmingham; Pediatric Nephrology, Birmingham, Alabama
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Providence Clinical Research, Burbank, California
  - AIDS Research Alliance, Los Angeles, California
  - UCLA Medical center Medicine/Nephrology, Los Angeles, California
  - University of California Davis Health System, Sacramento, California
  - CALIFORNIA PACIFIC MEDICAL CENTER; Office of Dr. Venkat Peddi, San Francisco, California
  - University of Colorado; Kidney Transplant Center Office of Dr. Laurence Chan, Aurora, Colorado
  - New England Research Associates, Trumbull, Connecticut
  - Christiana Care Health System, Newark, Delaware
  - Omega Research Consultants, Orlando, Florida
  - Kendall South Medical Center Inc., South Miami, Florida
  - All Children'S Hospital; Pediatric Blood & Marrow Transplant Program, St. Petersburg, Florida
  - Vita Research Solutions, Inc, Tamarac, Florida
  - University of South Florida, Tampa, Florida
  - Piedmont Hospital; Transplant Services, Atlanta, Georgia
  - EMORY UNIVERSITY; Bone Marrow & Stem Cell Transplant Center, Atlanta, Georgia
  - Medical College of Georgia; Medicine/ Nephrology, Augusta, Georgia
  - Northwestern Memorial Hospital; Divison of Infectious Diseases/ Dept of Medicine, Chicago, Illinois
  - Rush Uni Medical Center; Medicine/ Section of Infectious Diseases, Chicago, Illinois
  - University of Chicago; Infectious Disease, Chicago, Illinois
  - Tulane University Medical Center, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Brigham & Women'S Hospital, Boston, Massachusetts
  - Western New England Renal & Transplant Associates, P.C., Springfield, Massachusetts
  - Uni of Michigan Medical Center; Internal Medicine/ Infectious Disease, Ann Arbor, Michigan
  - Karmanos Cancer Inst. ; Hudson Webber; Cancer Research Building, Detroit, Michigan
  - Henry Ford Health System; Gastroenterology, Detroit, Michigan
  - Wayne State University School of Medicine, Detroit, Michigan
  - Beals Institute PC, Lansing, Michigan
  - Washington University; Wash Uni. Sch. Of Med, St Louis, Missouri
  - Our Lady of Lourdes Medical Center; Transplant Dept, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Long Island Jewish/North Shore Hospital, New Hyde Park, New York
  - Mount Sinai Medical Center; Division of Liver Diseases, New York, New York
  - DJL Clinical Research PLLC, Charlotte, North Carolina
  - Novant Health Pulmonary and Critical Care, Matthews, North Carolina
  - Duke University Health Systems, Raleigh, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Uni of Cincinnati Medical Center; Nephrology & Hypertension, Cincinnati, Ohio
  - Cleveland Clinic Foundation; Infectious Disease, Cleveland, Ohio
  - Toledo Hospital, Toledo, Ohio
  - Nazih Zuhdi Transplant Inst. ; Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University; College of Medicine, Philadelphia, Pennsylvania
  - Uni of Pennsylvania; Infectious Diseases, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Children'S Hospital of Pittsburgh; Infectious Disease, Pittsburgh, Pennsylvania
  - Medical University of South Carolina; Pediatric Cardiology, Charleston, South Carolina
  - Children'S Medical Center of Dallas, Dallas, Texas
  - Baylor University Medical Center Transplant Administration, Dallas, Texas
  - UT Southwestern Medical Center; Pediatrics Dept., Dallas, Texas
  - Sammons Cancer Center-Baylor University; Blood & Marrow Transplantation, Dallas, Texas
  - The Methodist Hospital, Houston, Texas
  - M.D Anderson Cancer Center; Infectious Diseases, Infection Control, and Employee Health, Houston, Texas
  - Texas Tech University Health Sciences Center; Department of Urology, Lubbock, Texas
  - University of Texas Health Science Center Transplant center, San Antonio, Texas
  - Scott and White Division of Nephrology Dept of Medicine, Temple, Texas
  - University of Utah Health Science Center Gastroenterology, Salt Lake City, Utah
- Argentina (6):
  - Hospital General de Agudos Juan Antonio Fernandez; infectología, Buenos Aires
  - Instituto Medico Platense, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma Buenos Aires
  - Hospital General de Agudos Dr. Ignacio Pirovano, Ciudad Autonoma Buenos Aires
  - Hospital Italiano de La Plata, La Plata
  - Hospital de Niños Dr. Orlando Alassia, Santa Fe
- Belgium (4):
  - Onze Lieve Vrouwziekenhuis Aalst, Aalst
  - Institut Jules Bordet, Brussels
  - Hospital Erasme; Neurologie, Brussels
  - UZ Brussel, Brussels
- Brazil (5):
  - Fiocruz - Fundação Oswaldo Cruz, Rio de Janeiro, Rio de Janeiro
  - Hospital Alemao Oswaldo Cruz; Oncologia, São Paulo, São Paulo
  - Iop - Graacc - Unifesp, São Paulo, São Paulo
  - Hospital do Rim e Hipertensão - Fundação Oswaldo Ramos, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Bulgaria (4):
  - UMHA - Sv. Georgi; Clinic of Nephrology & Haemodialysis, Plovdiv
  - UMHAT Sv. Georgi, EAD; Clinic of Infectious Diseases, Plovdiv
  - Mhat Alexandrovska Ead ; Clinic of Nephrology & Transplantation, Uni Hospital, Sofia
  - Specialized Hospital for children with oncohaematologica Diseases; Dept. Of Transplantations, Sofia
- Canada (2):
  - Uni of Manitoba; Faculty of Medicine, Winnipeg, Manitoba
  - St Paul'S, Saskatoon, Saskatchewan
- Chile (3):
  - Hospital Luis Calvo Mackenna; Unidad de Investigacion, Santiago
  - Hospital Dr. Sotero del Rio, Santiago
  - Centro de Investigaciones Clinicas Viña del Mar, Viña Del Mar Valparaiso
- Colombia (4):
  - Infectologos Asociados, Barranquilla
  - Simedics Ips, Bogotá
  - Centro de Investigaciones Clinicas S.A.S, Cali
  - Fundacion Cardiovascular de Colombia - Instituto del Corazón, Floridablanca
- Czechia (7):
  - Fakultni nemocnice Brno; Interni hematologicka a onkologicka klinika, Brno
  - Fakultni Nemocnice; Hemato-Oncology, Pilsen
  - The Institute of Hematology and Blood Transfusion Transplantation Unit; Hematology and Blood Transf, Prague
  - Fakultni nemocnice v Motole; Klinika detske hematologie a onkologie UK 2.LF, Prague
  - KASMED, s.r.o.; Alergologie a klinicka imunologie, Tábor
  - Revmatologicka Ambulance-Terezin, Terezín
  - Revmatologicka ambulance, Zlín
- Estonia (5):
  - West Tallinn Central Hospital; Nephrology, Tallinn
  - North Estonia medical Centre; Hematology, Tallinn
  - Tartu Uni Clinics; Clinic of Surgery & Internal Medicine Dept of Nephrology, Tartu
  - Tartu Uni Hospital; Hematology - Oncology Clinic, Tartu
  - Tartu University Hospital; Department of Infectious Diseases, Tartu
- France (6):
  - Centre Hospitalier de la Croix Rousse, Lyon
  - Hopital Robert Debre; Pediatric Hematology Dept, Paris
  - Hopital Saint Louis; Service de Nephrologie - Transplantation, Paris
  - Hopital Europeen Georges Pompidou; Service de Nephrologie, Paris
  - Hopital Rangueil; Nephrologie, Toulouse
  - CHRU Bretonneau, Tours
- Germany (8):
  - Uniklinik RWTH Aachen; Med. Klinik II; Klinik für Nephrologie und klinische Immunologie, Aachen
  - Charite - Campus Virchow Klinikum; Abteilung fuer Chirurgie, Berlin
  - Universitätsklinikum Essen; Innere Klinik und Poliklinik für Tumorforschung, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - UNI-Klinikum Heidelberg Chirurgische Klinik, Heidelberg
  - Ludwig-Maximilian-Universitaetsklinik; Med. Poliklinik/Infektiologie, München
  - Ludwig-Maximilians-Universitaet; Medizinische Klinik und Poliklinik IV, München
  - Universitaetsklinikum Muenster; Paedriatrische Haematologie und Onkologie, Münster
- Guatemala (5):
  - Clinica Familiar Luis Angel Garcia, Guatemala City
  - CERICAP, Guatemala City
  - Centro de Investigaciones Pediatricas, Guatemala City
  - Hospital Roosevelt Guatemala; Clinica de Infecciosas, Guatemala City
  - Unidad Nacional de Oncologia Pediatrica, Guatemala City
- Hungary (10):
  - Fov.Onk.Egyesitett Szt. Istvan es Szt Laszlo Korh.-Rend.Int., Budapest
  - Debreceni Egyetem, Orvos- és Egészségtudományi Centrum;, Debrecen
  - Petz Aladar Megyei Korhaz; Hematologia, Győr
  - Bekes Megyei Kepviselotestulet Pandy Kalman Korhaza, Gyula
  - Békés Megyei Pándy Kálmán Kórház; Onkologiai tanszek, Gyula
  - Pecsi Tudomanyegyetem, Pécs
  - University of Szeged; Transplantation Department, Szeged
  - Fejer Megyei Szent Gyorgy Korhaz, Székesfehérvár
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rend.Int., Szolnok
  - Veszprem Megyei Csolnoky Ferenc Korhaz Nonprofit Zrt., Veszprém
- Israel (8):
  - Rambam Health Care Campus; Hematology, Haifa
  - Hadassah University Hospital - Ein Kerem; BMT & Cancer Immunotherapy Dept., Jerusalem
  - Rabin MC- Belinson campus, Petah Tikva
  - Rabin Medical Center-Golda Campus - Hasharon; Department of Transplantation, Petah Tikva
  - Rabin Medical Center; Liver Inst., Petah Tikva
  - Chaim Sheba Medical Center; Hematology BMT & CBB, Ramat Gan
  - Sourasky MC; Transplant Unit, Tel Aviv
  - Chaim Sheba MC; Pediatric Hematology Oncology, Tel Litwinsky
- Italy (7):
  - Azienda Ospedaliera; Divisione Malattie Infettive E Tropicali, Parma, Emilia-Romagna
  - POLICLINICO Universitatio A.Gemelli, Div. Chirurgia Generale e Trapianti d'Organo, Rome, Lazio
  - I.N.M.I. L. Spallanzani IRCCS, Rome, Lazio
  - ASST DEGLI SPEDALI CIVILI DI BRESCIA; Dipartimento Malattie Infettive, Brescia, Lombardy
  - ASST DI MONZA; Divisione Malattie Infettive, Monza, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico; Clinica Pediatica De Macchi, Milano, Molise
- Latvia (2):
  - Latvia Transplantation Center P. Stradina Hospital; Transplantation, Riga
  - Children's Clinical University Hospital, Riga
- Lithuania (6):
  - Kaunas Clinics Public Institution; Clinic of Nephrology, Kaunas
  - Klaipeda University Hospital; Public Institution, Klaipėda
  - Siauliai Republican Hospital Public Institution, Šiauliai
  - Vilnius University Hospital Santariskiu Clinic, Hematology, Oncology and Tranfusion Medicine Center, Vilnius
  - Vilnius University Hospital Santariskiu Clinic, Vilnius
  - Republican Tuberculosis and Infectious Diseases University H, Vilnius
- Mexico (7):
  - Phylaxis Clinical Research S de RL de CV, Cuautitlán Izcalli
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde; Infectología piso 7, Guadalajara
  - Centro de Investigacion Clínica GRAMEL S.C, México
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador; Infectologia, México
  - INER- Instituto Nacional de Enfermedades Respiratorias"Ismae, México
  - Hospital Universitario de Monterrey; Infectologia, Monterrey
  - Hospital de Especialidades del Centro Medico Puerta de Hierr, Zapopan
- Poland (10):
  - Wojewodzki Szp.Specjalistyczny im.K.Dluskiego w Bialymstoku, Bialystok
  - NZOZ Vitamed, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - SPZOZ Szpital Uniw W Krakowie, Krakow
  - SPZOZ Uniwersytecki Szp Klin; nr1 im.N.Barlickiego UM, Lodz
  - SPSK nr 2 Pomorskiej Akademii Medycznej w Szczecinie, Szczecin
  - Szpital Dzieciatka Jezus-Centrum Lecezenia Obrazen; Dpt of Transplantation Medicine & Nephrology, Warsaw
  - Instytut Pomnik-Centrum Zdrowia Dziecka, Klinika Nefrologii, Transp. Nerek i Nadcisnienia Tetniczego, Warsaw
  - SP Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw
  - ALL-MED Specjalistyczna Opieka Medyczna, Wroclaw
- Institutul de Urologie Si Transplant Renal Fundeni, Bucharest, Romania
- South Africa (17):
  - Josha Research, Bloemfontein
  - Londisizwe Research Centre, Durban
  - Sebastian Peter, Durban
  - Dr V Naidoo Private Practice, Durban
  - Govind U, Durban
  - Soweto CTC - Dr Phoshoko site, Johannesburg
  - Soweto CTC - Dr Mushwana site, Johannesburg
  - Newtown Clinical Research, Johannesburg
  - Mzansi Ethical Research Centre, Middelburg
  - Be Part Yoluntu Centre, Paarl
  - Global Clinical Trials Port Elizabeth, Port Elizabeth
  - Kalafong Hospital; Pathology, Pretoria
  - Emmed Research, Pretoria
  - Synexus Clinical Research Centres SA Stanza Bopape, Pretoria
  - Soweto Clinical Trial Centre, Soweto
  - Tygerberg Hospital Pediatrics and Child Health, Tygerberg; Cape Town
  - Welkom Clinical Trial Centre, Welkom
- Spain (13):
  - Hospital Universitari de Bellvitge; Servicio de Nefrologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, LA Coruña
  - Hospital Universitari Vall d'Hebron; Departamento de Enfermedades Infecciosas, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Clinico San Carlos; Servicio de Nefrologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Enfermedades Infecciosas, Madrid
  - Hospital Universitario 12 de Octubre; HIV Unit, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Pediatria, Madrid
  - Hospital Universitario La Paz; Hepatología y Trasplantes, Madrid
  - Hospital Universitario la Paz; Servicio de Enfermedades Infecciosas - HIV unit, Madrid
- Universitätsspital Zürich; Klinik für Nephrologie, Zurich, Switzerland
- Ukraine (4):
  - Ukrainian Pediatric Specialized Hospital of Ministry of Health of Ukraine Dept of BMT, Kiev
  - Institute of Nephrology AMS; Dept of Nephrology & dialysis, Kiev
  - Lugansk Regional Clinical Hospital; Chair of Therapy Faculty of Postgr.Ed, Lugnansk
  - Zaporozhye State Medical University; Dept of Transplantology, Zaporizhzhya
- United Kingdom (3):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Manchester Royal Infirmary; Renal Transplant Unit, Manchester
  - Nottingham City Hospital; Transplant Unit, Nottingham

REFERENCES:
- [Derived] Mitha E, Krivan G, Jacobs F, Nagler A, Alrabaa S, Mykietiuk A, Kenwright A, Le Pogam S, Clinch B, Vareikiene L. Safety, Resistance, and Efficacy Results from a Phase IIIb Study of Conventional- and Double-Dose Oseltamivir Regimens for Treatment of Influenza in Immunocompromised Patients. Infect Dis Ther. 2019 Dec;8(4):613-626. doi: 10.1007/s40121-019-00271-8. Epub 2019 Oct 30. PMID 31667696

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow is provided for the safety analysis population, which was the primary analysis population for evaluation of safety. Safety population included all participants who received at least one dose of study drug and had a safety assessment performed post randomization. Participants were reported under the actual treatment received.
Groups:
- Conventional Dose: Immunocompromised participants received oseltamivir syrup at a dose ranging from 30 to 75 mg based on body weight, twice daily for children (1 to 12 years old) and oseltamivir capsules 75 mg twice daily for adults/adolescents greater than or equal to (>/=) 13 years old or placebo-matched to oseltamivir twice daily over 10 days.
- Double Dose: Immunocompromised participants received oseltamivir syrup at a dose ranging from 60 to 150 mg based on body weight, twice daily for children (1 to 12 years old) and oseltamivir capsules 150 mg twice daily for adults/adolescents (>/=13 years old) or placebo matched to oseltamivir twice daily over 10 days.
Period: Overall Study
Arm/Group | Conventional Dose | Double Dose
Started | 105 | 110
Completed | 99 | 100
Not Completed | 6 | 10
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 5 | 6
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Dose | Double Dose | Total
Number analyzed (Participants) | 105 | 110 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (15.5) | 43.9 (16.5) | 43.5 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 62 | 119
  Male | 48 | 48 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 21 | 36
  Not Hispanic or Latino | 90 | 89 | 179
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 3 | 9
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 33 | 60
  White | 72 | 72 | 144
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to Day 40
Population: The safety population included all participants who received at least one dose of study drug and had a safety assessment performed post randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 105 | 110
percentage of participants
  On Treatment | 40.0 | 47.3
  Off Treatment | 25.7 | 29.1

2. Primary Outcome: Percentage of Participants Who Developed Viral Resistance to Oseltamivir
Description: Resistance was defined as the presence of oseltamivir resistance mutations in viruses isolated from nasopharyngeal swab samples, identified by sequencing of the neuraminidase (NA) and hemagglutinin (HA) genes (genotypic resistance) and/or determination of the oseltamivir concentration at which the response is reduced by half (IC50) in an NA inhibition assay (phenotypic resistance). Reported are post-baseline phenotypic and genotypic resistance in adults >/= 18 years and children and adolescents <18 years in the modified Intent-to-Treat infected (mITTi) population.
Time Frame: Baseline up to Day 40
Population: mITTi population: all participants randomized to a particular treatment, regardless of whether they received that treatment or not, who received at least one dose of study drug and with central laboratory confirmation of influenza infection, excluding participants infected with oseltamivir-resistant influenza at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 81 | 86
percentage of participants
  Post-BL Phenotypic Resist, >/= 18 years: number analyzed (Participants) | 73 | 78
  Post-BL Phenotypic Resist, >/= 18 years | 8.2 | 1.3
  Post-BL Genotypic Resist, >/= 18 years: number analyzed (Participants) | 73 | 78
  Post-BL Genotypic Resist, >/= 18 years | 9.6 | 2.6
  Post-BL Phenotypic Resist, < 18 years: number analyzed (Participants) | 8 | 8
  Post-BL Phenotypic Resist, < 18 years | 25.0 | 0
  Post-BL Genotypic Resist, < 18 years: number analyzed (Participants) | 8 | 8
  Post-BL Genotypic Resist, < 18 years | 25.0 | 12.5

3. Primary Outcome: Percentage of Participants With Tissue Rejection or Graft Versus Host Disease (GVHD)
Description: The percentage of transplant patients in the safety population who experienced tissue rejection and/or GvHD is reported.
Time Frame: Baseline up to Day 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 105 | 110
percentage of participants | 0 | 0

4. Secondary Outcome: Time to Resolution (TTR) of All Clinical Influenza Symptoms
Description: TTR of all clinical influenza symptoms was defined as the time from treatment initiation to the start of the 24-hour period in which all 7 influenza symptoms had scores </= 1 (mild) and remained </=1 for at least 21.5 hours. . Reported are TTRs in adults >/= 18 years, adults and adolescents >/= 13 years and children <13 years in the mITTi population.
Time Frame: Baseline up to Day 40
Population: mITTi: all participants randomized to a particular treatment, regardless of whether they received that treatment or not, who received at least one dose of study drug and with central laboratory confirmation of influenza infection, excluding participants infected with oseltamivir-resistant influenza at baseline, and for whom data were available.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 82 | 86
hours
  Adults >/= 18 years: number analyzed (Participants) | 71 | 75
  Adults >/= 18 years | 103.3 [69.0 to 112.7] | 103.6 [57.1 to 140.0]
  Adults and adolescents >/= 13 years: number analyzed (Participants) | 75 | 78
  Adults and adolescents >/= 13 years | 103.4 [75.4 to 122.7] | 107.2 [63.9 to 140.0]
  Children < 13 years: number analyzed (Participants) | 4 | 5
  Children < 13 years | 32.1 [20.2 to NA] — Not Available due to insufficient number of data points. | 115.9 [45.5 to 495.0]

5. Secondary Outcome: Total Symptom Score Area Under the Efficacy Curve (AUE)
Description: The overall extent and severity of illness was quantified by the AUE of the total symptom scores over the duration of illness, i.e., from the start of treatment to the time symptoms first alleviated. Total symptom scores were calculated from the sum of seven individual symptom scores with each individual symptom scored from 0 (healthy) to 3 (worst sickness) and a maximum total symptom score of 21. The AUE of these average scores was then calculated for each participant using the trapezoidal rule (the trapezoidal rule calculates the area under any curve by adding up all trapezoids under such a curve). A larger area indicates more severe disease. In this study participants were treated for 10 days. If a participant had scored 21 on every visit then AUE would have been 21 score x 10 days x 24 hours/day =5040 score x hours units, which is the highest possible score. The lowest possible score is 0. Reported are results for adults >/= 18 years in the mITTi population.
Time Frame: Baseline up to Day 40
Population: as for outcome 2
Measure: Median (Full Range); unit: score * hour
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 59 | 67
score * hour | 774.7 [60.8 to 11435.5] | 811.5 [63.0 to 8648.1]

6. Secondary Outcome: Time to Resolution of Fever
Description: Fever was defined as temperature >/= 37.8 degrees Celsius at any time point during the study. TTR of fever was determined in Adults >/= 18 years, Adults and adolescents >/= 13 years and Children < 13 years of the mITTi population.
Time Frame: Baseline up to Day 40
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 38 | 35
hours
  Adults >/= 18 years: number analyzed (Participants) | 35 | 32
  Adults >/= 18 years | 11.0 [0.0 to 16.2] | 0.5 [0.0 to 8.8]
  Adults and adolescents >/= 13 years: number analyzed (Participants) | 37 | 33
  Adults and adolescents >/= 13 years | 11.0 [0.0 to 16.2] | 0.5 [0.0 to 8.8]
  Children < 13 years: number analyzed (Participants) | 1 | 2
  Children < 13 years | NA [NA to NA] — Not Available: participant censored for analysis | 26.0 [NA to NA] — CI not available for only 2 participants: actual measure values for these participants were 0.0 and 51.9.

7. Secondary Outcome: Change From Baseline in Viral Load Assessed by Culture
Description: Nasopharyngeal swab samples were cultured in Madin-Darby Canine Kidney cells. Culture supernatants were harvested after 2 weeks, or after a full-blown cytopathic effect was observed. Presence of infectious viruses in the cell culture supernatants (viral titer), expressed as log10 50% Tissue Culture Infectious Dose/milliliter (TCID50/mL), was determined by hemagglutination assay using turkey erythrocytes for H1 and B viruses or by detection of the virus nucleoprotein (NP) using ELISA for H3 viruses. A value of < 0.5 log10 TCID50/mL was interpreted as negative. Data are reported for adults >/= 18 years and adolescents and children < 18 years.
Time Frame: Baseline (Day 1), Day 2/3, Day 6, Day 8, Day 11 end of treatment (EOT), follow-up (FU) Day 15 and FU Day 40.
Population: as for outcome 2
Measure: Median (Full Range); unit: TCID50/mL
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 81 | 86
TCID50/mL
  >/= 18 years, Baseline (BL): number analyzed (Participants) | 70 | 76
  >/= 18 years, Baseline (BL) | 3.38 [0.5 to 6.0] | 3.75 [0.5 to 6.3]
  >/= 18 years, Change from BL on Day 2/3: number analyzed (Participants) | 67 | 73
  >/= 18 years, Change from BL on Day 2/3 | -1.50 [-5.3 to 0.8] | -1.50 [-5.0 to 1.50]
  >/= 18 years, Change from BL on Day 6: number analyzed (Participants) | 65 | 71
  >/= 18 years, Change from BL on Day 6 | -2.50 [-5.5 to 0.0] | -3.00 [-5.8 to 1.0]
  >/= 18 years, Change from BL on Day 8: number analyzed (Participants) | 62 | 62
  >/= 18 years, Change from BL on Day 8 | -2.75 [-5.5 to 0.0] | -3.25 [-5.8 to 0.0]
  >/= 18 years, Change from BL on Day 11: number analyzed (Participants) | 64 | 71
  >/= 18 years, Change from BL on Day 11 | -2.88 [-5.5 to 0.0] | -3.25 [-5.8 to 0.3]
  >/= 18 years, Change from BL on Day 15: number analyzed (Participants) | 62 | 65
  >/= 18 years, Change from BL on Day 15 | -3.00 [-5.5 to 0.3] | -3.25 [-5.8 to 0.0]
  >/= 18 years, Change from BL on Day 40: number analyzed (Participants) | 64 | 65
  >/= 18 years, Change from BL on Day 40 | -3.00 [-5.5 to 0.0] | -3.25 [-5.8 to 0.0]
  < 18 years, BL: number analyzed (Participants) | 8 | 8
  < 18 years, BL | 3.13 [0.8 to 6.0] | 4.00 [1.8 to 5.3]
  < 18 years, Change from BL on Day 2/3: number analyzed (Participants) | 7 | 8
  < 18 years, Change from BL on Day 2/3 | -1.00 [-2.3 to 0.8] | -2.00 [-3.3 to 0.0]
  < 18 years, Change from BL on Day 6: number analyzed (Participants) | 7 | 7
  < 18 years, Change from BL on Day 6 | -2.00 [-3.3 to -0.3] | -3.50 [-4.8 to -2.3]
  < 18 years, Change from BL on Day 8: number analyzed (Participants) | 5 | 7
  < 18 years, Change from BL on Day 8 | -2.50 [-3.3 to -0.3] | -3.50 [-4.8 to -1.3]
  < 18 years, Change from BL on Day 11: number analyzed (Participants) | 7 | 7
  < 18 years, Change from BL on Day 11 | -2.50 [-5.3 to 0.0] | -3.50 [-4.8 to -2.3]
  < 18 years, Change from BL on Day 15: number analyzed (Participants) | 7 | 7
  < 18 years, Change from BL on Day 15 | -2.50 [-5.3 to 1.0] | -3.50 [-4.8 to -2.3]
  < 18 years, Change from BL on Day 40: number analyzed (Participants) | 7 | 8
  < 18 years, Change from BL on Day 40 | -2.50 [-5.3 to 0.3] | -3.50 [-4.8 to -1.3]

8. Secondary Outcome: Percentage of Participants With Viral Shedding Assessed by Culture Over Time
Description: Viral shedding was determined through measurement of the viral titer after viral culture in Madin-Darby Canine Kidney cells by hemagglutination assay (for Flu A/H1N1 and Flu B) and NP-ELISA (for Flu A/H3N2) and expressed in log10 TCID50/mL. Reported is the percentage of participants with viral shedding over time in adults >/= 18 years and adolescents and children < 18 years.
Time Frame: Baseline (Day 1), Day 2/3, Day 6, Day 8, Day 11 end of treatment (EOT), follow-up (FU) Day 15 and FU Day 40.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 81 | 86
percentage of participants
  >/= 18 years, Baseline: number analyzed (Participants) | 70 | 76
  >/= 18 years, Baseline | 91.4 | 84.2
  >/= 18 years, Day 2/3: number analyzed (Participants) | 67 | 73
  >/= 18 years, Day 2/3 | 67.2 | 58.9
  >/= 18 years, Day 6: number analyzed (Participants) | 65 | 71
  >/= 18 years, Day 6 | 15.4 | 18.3
  >/= 18 years, Day 8: number analyzed (Participants) | 63 | 62
  >/= 18 years, Day 8 | 3.2 | 4.8
  >/= 18 years, Day 11: number analyzed (Participants) | 65 | 71
  >/= 18 years, Day 11 | 1.5 | 4.2
  >/= 18 years, Day 15: number analyzed (Participants) | 63 | 65
  >/= 18 years, Day 15 | 7.9 | 1.5
  >/= 18 years, Day 40: number analyzed (Participants) | 65 | 65
  >/= 18 years, Day 40 | 0.0 | 0.0
  < 18 years, Baseline: number analyzed (Participants) | 8 | 8
  < 18 years, Baseline | 100.0 | 100.0
  < 18 years, Day 2/3: number analyzed (Participants) | 7 | 8
  < 18 years, Day 2/3 | 71.4 | 75.0
  < 18 years, Day 6: number analyzed (Participants) | 7 | 7
  < 18 years, Day 6 | 42.9 | 0.0
  < 18 years, Day 8: number analyzed (Participants) | 5 | 7
  < 18 years, Day 8 | 0.0 | 0.0
  < 18 years, Day 11: number analyzed (Participants) | 7 | 7
  < 18 years, Day 11 | 14.3 | 0.0
  < 18 years, Day 15: number analyzed (Participants) | 7 | 7
  < 18 years, Day 15 | 28.6 | 0.0
  < 18 years, Day 40: number analyzed (Participants) | 7 | 8
  < 18 years, Day 40 | 0.0 | 0.0

9. Secondary Outcome: Time to Cessation of Viral Shedding by Cell Culture
Description: Viral shedding was determined through measurement of the viral titer after viral culture in Madin-Darby Canine Kidney cells by hemagglutination assay (for Flu A/H1N1 and Flu B) and NP-ELISA (for Flu A/H3N2) and expressed in log10 TCID50/mL. Reported is the time to cessation of viral shedding over time in adults >/= 18 years and adolescents and children < 18 years.
Time Frame: Baseline up to Day 40
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 81 | 86
hours
  >/= 18 years: number analyzed (Participants) | 64 | 64
  >/= 18 years | 105.0 [98.3 to 109.2] | 105.4 [83.0 to 107.7]
  < 18 years: number analyzed (Participants) | 8 | 8
  < 18 years | 150.3 [34.2 to 891.3] | 94.9 [8.6 to 109.4]

10. Secondary Outcome: Change From Baseline in Viral Load Assessed by Reverse Transcription Polymerase Chain Reaction (RT-PCR)
Description: Nasopharyngeal swab samples were tested for influenza A and B RNA using semi-quantitative RT-PCR specific for influenza A and B matrix gene, respectively, after viral RNA isolation. Cycle threshold (Ct) value was determined for each sample. Conversion of Ct values into viral load, expressed as log10 virus particles/mL (vp/mL), was obtained using external standard curves ran in parallel in all RT-PCR experiments. A value of < 2.6 log10 vp/mL for Flu A strains and < 3.0 log10 vp/mL for Flu B strains was interpreted as a negative result. Data are reported for adults >/= 18 years and adolescents and children < 18 years.
Time Frame: Baseline (Day 1), Day 2/3, Day 6, Day 8, Day 11 end of treatment (EOT), follow-up (FU) Day 15 and FU Day 40.
Population: as for outcome 2
Measure: Median (Full Range); unit: log10 vp/mL
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 81 | 86
log10 vp/mL
  >/= 18 years, Baseline (BL): number analyzed (Participants) | 72 | 76
  >/= 18 years, Baseline (BL) | 6.47 [2.7 to 8.8] | 6.52 [2.8 to 8.5]
  >/= 18 years, Change from BL on Day 2/3: number analyzed (Participants) | 65 | 67
  >/= 18 years, Change from BL on Day 2/3 | -1.20 [-6.4 to 1.6] | -1.35 [-4.6 to 1.1]
  >/= 18 years, Change from BL on Day 6: number analyzed (Participants) | 41 | 39
  >/= 18 years, Change from BL on Day 6 | -2.36 [-8.0 to 0.1] | -2.34 [-7.7 to 0.1]
  >/= 18 years, Change from BL on Day 8: number analyzed (Participants) | 28 | 20
  >/= 18 years, Change from BL on Day 8 | -2.66 [-5.4 to -0.3] | -2.62 [-7.8 to -0.3]
  >/= 18 years, Change from BL on Day 11: number analyzed (Participants) | 19 | 17
  >/= 18 years, Change from BL on Day 11 | -3.51 [-7.3 to -2.2] | -2.96 [-4.5 to 1.3]
  >/= 18 years, Change from BL on Day 15: number analyzed (Participants) | 10 | 6
  >/= 18 years, Change from BL on Day 15 | -3.63 [-8.0 to -0.9] | -2.60 [-3.4 to 0.0]
  >/= 18 years, Change from BL on Day 40: number analyzed (Participants) | 3 | 1
  >/= 18 years, Change from BL on Day 40 | -4.80 [-5.4 to 0.8] | -7.71 [-7.71 to -7.71]
  < 18 years, BL: number analyzed (Participants) | 8 | 8
  < 18 years, BL | 5.88 [2.8 to 7.7] | 5.96 [5.5 to 7.3]
  < 18 years, Change from BL on Day 2/3: number analyzed (Participants) | 6 | 8
  < 18 years, Change from BL on Day 2/3 | -0.66 [-2.7 to 1.4] | -0.71 [-5.6 to 0.4]
  < 18 years, Change from BL on Day 6: number analyzed (Participants) | 6 | 4
  < 18 years, Change from BL on Day 6 | -1.97 [-2.7 to 0.3] | -1.73 [-2.7 to -1.2]
  < 18 years, Change from BL on Day 8: number analyzed (Participants) | 1 | 3
  < 18 years, Change from BL on Day 8 | 1.56 [1.56 to 1.56] | -2.26 [-2.9 to -1.5]
  < 18 years, Change from BL on Day 11: number analyzed (Participants) | 2 | 1
  < 18 years, Change from BL on Day 11 | -0.89 [-3.2 to 1.4] | -2.41 [-2.41 to -2.41]
  < 18 years, Change from BL on Day 15: number analyzed (Participants) | 3 | 0
  < 18 years, Change from BL on Day 15 | 1.26 [-2.9 to 1.9] |

11. Secondary Outcome: Percentage of Participants With Viral Shedding Assessed by RT-PCR Over Time
Description: Viral shedding was determined by direct viral load measurement from nasopharyngeal swabs by RT-PCR assay and expressed in log10 vp/mL. Reported is the percentage of subjects with viral shedding over time in adults >/= 18 years and adolescents and children < 18 years.
Time Frame: Baseline (Day 1), Day 2/3, Day 6, Day 8, Day 11 end of treatment (EOT), follow-up (FU) Day 15 and FU Day 40.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 81 | 86
percentage of participants
  >/= 18 years, Baseline: number analyzed (Participants) | 72 | 78
  >/= 18 years, Baseline | 100.0 | 97.4
  >/= 18 years, Day 2/3: number analyzed (Participants) | 69 | 75
  >/= 18 years, Day 2/3 | 92.8 | 88.0
  >/= 18 years, Day 6: number analyzed (Participants) | 67 | 73
  >/= 18 years, Day 6 | 56.7 | 49.3
  >/= 18 years, Day 8: number analyzed (Participants) | 65 | 64
  >/= 18 years, Day 8 | 41.5 | 23.4
  >/= 18 years, Day 11: number analyzed (Participants) | 67 | 73
  >/= 18 years, Day 11 | 25.4 | 21.9
  >/= 18 years, Day 15: number analyzed (Participants) | 66 | 67
  >/= 18 years, Day 15 | 10.6 | 9.0
  >/= 18 years, Day 40: number analyzed (Participants) | 68 | 67
  >/= 18 years, Day 40 | 1.5 | 1.5
  < 18 years, Baseline: number analyzed (Participants) | 8 | 8
  < 18 years, Baseline | 100.0 | 100.0
  < 18 years, Day 2/3: number analyzed (Participants) | 7 | 8
  < 18 years, Day 2/3 | 85.7 | 75.0
  < 18 years, Day 6: number analyzed (Participants) | 7 | 7
  < 18 years, Day 6 | 85.7 | 57.1
  < 18 years, Day 8: number analyzed (Participants) | 5 | 7
  < 18 years, Day 8 | 20.0 | 42.9
  < 18 years, Day 11: number analyzed (Participants) | 7 | 7
  < 18 years, Day 11 | 28.6 | 14.3
  < 18 years, Day 15: number analyzed (Participants) | 7 | 7
  < 18 years, Day 15 | 42.9 | 0.0
  < 18 years, Day 40: number analyzed (Participants) | 7 | 8
  < 18 years, Day 40 | 0.0 | 0.0

12. Secondary Outcome: Time to Cessation of Viral Shedding by RT-PCR
Description: Viral shedding was determined by direct viral load measurement from nasopharyngeal swabs by RT-PCR assay and expressed in log10 vp/mL. Reported is the time to cessation of viral shedding over time in adults >/= 18 years and adolescents and children < 18 years.
Time Frame: Baseline up to Day 40
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 81 | 86
hours
  >/= 18 years: number analyzed (Participants) | 72 | 76
  >/= 18 years | 178.0 [152.2 to 227.0] | 154.1 [128.5 to 171.0]
  < 18 years: number analyzed (Participants) | 8 | 8
  < 18 years | 181.0 [106.2 to 943.7] | 180.5 [8.6 to 247.8]

13. Secondary Outcome: Percentage of Participants With Persistent Viral Shedding
Description: Persistent shedding was defined as a viral load reduction <1 log10 vp/mL at end of treatment compared with baseline. Reported is the percentage of participants with persistent viral shedding at end of treatment in adults >/= 18 years and adolescents and children < 18 years.
Time Frame: Baseline to Day 11 (EOT)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 81 | 86
percentage of participants | 1.2 | 4.7

14. Secondary Outcome: Percentage of Participants Who Developed Secondary Illness
Description: Secondary illness included bronchitis, pneumonia, acute sinusitis, sinusitis, lower respiratory infection or otitis media. Reported is the percentage of participants with at least one event in adults >/= 18 years and adolescents and children < 18 years.
Time Frame: Baseline up to Day 40
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 81 | 86
percentage of participants
  >/=18 years: number analyzed (Participants) | 73 | 78
  >/=18 years | 8.2 | 5.1
  < 18 years: number analyzed (Participants) | 8 | 8
  < 18 years | 12.5 | 0.0

15. Secondary Outcome: Percentage of Participants Who Initiated Antibiotic Treatment
Description: Secondary illness included bronchitis, pneumonia, acute sinusitis, sinusitis, lower respiratory infection or otitis media. Reported is the percentage of participants with secondary illness, who initiated antibiotic treatment, in adults >/= 18 years and adolescents and children < 18 years.
Time Frame: Baseline up to Day 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 105 | 110
percentage of participants
  >/= 18 years: number analyzed (Participants) | 98 | 101
  >/= 18 years | 8.2 | 5.0
  < 18 years: number analyzed (Participants) | 7 | 9
  < 18 years | 14.3 | 0.0

16. Secondary Outcome: Percentage of Participants Hospitalized
Description: Reported is the percentage of participants, who required hospitalization at any time between treatment initiation and the end of the study period, in adults >/= 18 years and adolescents and children < 18 years.
Time Frame: Baseline up to Day 40
Population: The ITTi population included all participants randomized and with central laboratory confirmation of influenza infection, excluding participants infected with oseltamivir-resistant influenza at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 83 | 86
percentage of participants
  >/= 18 years: number analyzed (Participants) | 74 | 78
  >/= 18 years | 6.8 | 7.7
  < 18 years: number analyzed (Participants) | 9 | 8
  < 18 years | 11.1 | 0.0

17. Secondary Outcome: Duration of Hospitalization
Description: Reported is the duration of hospitalization at any time between treatment initiation and the end of the study period, in adults >/= 18 years and adolescents and children < 18 years.
Time Frame: Baseline up to Day 40
Population: as for outcome 16
Measure: Median (Full Range); unit: days
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 83 | 86
days
  >/= 18 years: number analyzed (Participants) | 74 | 78
  >/= 18 years | 7.0 [5.0 to 14.0] | 6.50 [4.0 to 32.0]
  < 18 years: number analyzed (Participants) | 9 | 8
  < 18 years | 5.0 [5.0 to 5.0] | NA [NA to NA] — N/A=not available as no hospitalization occurred in this arm.

18. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of Oseltamivir in Adults
Description: Reported here are oseltamivir Cmax data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: The pharmacokinetic evaluable patient (PKEP) population comprised all participants in the ITT population who had at least one valid post-dose drug concentration measurement at a scheduled visit time point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
nanograms per milliliter (ng/mL) | 65.5 (26.8) | 149 (80.7)

19. Secondary Outcome: Pharmacokinetics: Trough Plasma Concentration (Ctrough) of Oseltamivir in Adults
Description: Reported here are oseltamivir Ctrough data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: The PKEP population comprised all participants in the ITT population who had at least one valid post-dose drug concentration measurement at a scheduled visit time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
ng/mL | 2.33 (0.641) | 6.98 (5.1)

20. Secondary Outcome: Pharmacokinetics : Area Under the Concentration-Time Curve From 0 to 12 Hours (AUC0-12) at Steady State of Oseltamivir in Adults
Description: AUC0-12 was reported at steady state as nanograms per hour per milliliter. (ng*hr/mL). Reported here are oseltamivir AUC0-12 data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
ng*hr/mL | 197 (49.7) | 501 (320)

21. Secondary Outcome: Pharmacokinetics: Time to Maximum Concentration (Tmax) of Oseltamivir in Adults
Description: Reported here are oseltamivir tmax data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
hour | 1.08 (0.484) | 1.08 (0.504)

22. Secondary Outcome: Pharmacokinetics: Elimination Constant (ke) of Oseltamivir in Adults
Description: Reported here are oseltamivir ke data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
1/hr | 5.15 (0.497) | 4.79 (1.25)

23. Secondary Outcome: Pharmacokinetics: Apparent Clearance (CL/F) of Oseltamivir in Adults
Description: Reported here are oseltamivir CL/F data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: liter/hour (L/hr)
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
liter/hour (L/hr) | 402 (96.0) | 367 (126)

24. Secondary Outcome: Pharmacokinetics: Apparent Volume of Distribution (Vc/F) of Oseltamivir in Adults
Description: Reported here are oseltamivir Vc/F data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: liter (L)
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
liter (L) | 77.5 (13.6) | 75.4 (17.5)

25. Secondary Outcome: Pharmacokinetics: Cmax of Oseltamivir Carboxylate in Adults
Description: Reported here are oseltamivir carboxylate Cmax data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
ng/mL | 655 (276) | 1420 (574)

26. Secondary Outcome: Pharmacokinetics: Ctrough of Oseltamivir Carboxylate in Adults
Description: Reported here are oseltamivir carboxylate Ctrough data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
ng/mL | 363 (167) | 831 (358)

27. Secondary Outcome: Pharmacokinetics : AUC0-12 at Steady State of Oseltamivir Carboxylate in Adults
Description: Reported here are oseltamivir carboxylate AUC0-12 data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: The PKEP population comprised all particiants in the ITT population who had at least one valid post-dose drug concentration measurement at a scheduled visit time point.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
ng*hr/mL | 6240 (2710) | 13800 (5670)

28. Secondary Outcome: Pharmacokinetics: Tmax of Oseltamivir Carboxylate in Adults
Description: Reported here are oseltamivir carboxylate tmax data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
hour | 3.83 (1.08) | 3.96 (0.841)

29. Secondary Outcome: Pharmacokinetics: Elimination Constant (ke) of Oseltamivir Carboxylate in Adults
Description: Reported here are oxeltamivir carboxylate ke data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
1/hr | 1.67 (0.681) | 1.61 (0.915)

30. Secondary Outcome: Pharmacokinetics: Apparent Clearance (CL/F) of Oseltamivir Carboxylate in Adults
Description: Reported here are oseltamivir carboxylate CL/F data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
L/hr | 14.0 (5.72) | 13.5 (7.66)

31. Secondary Outcome: Pharmacokinetics: Apparent Volume of Distribution (Vc/F) of Oseltamivir Carboxylate in Adults
Description: Reported here are oseltamivir carboxylate Vc/F data for adults >/= 18 years.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: liter (L)
Arm/Group | Conventional Dose | Double Dose
Number analyzed (Participants) | 9 | 13
liter (L) | 8.39 (0.00) | 8.39 (0.00)

32. Secondary Outcome: Pharmacokinetics: Cmax of Oseltamivir in Adolescents and Children
Description: Reported here are oseltamivir Cmax data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: ng/mL
Groups:
- Adolescents and Children With Pharmacokinetic Evaluation: This analysis set comprises participants < 18 years from both arms in the study who underwent pharmacokinetic evaluation. Immunocompromised participants in the Conventional dose arm received oseltamivir syrup at doses ranging from 30 to 75 mg based on body weight, twice daily for children (1 to 12 years old) and oseltamivir capsules 75 mg twice daily for adolescents greater than or equal to (>/=) 13 years old or placebo-matched to oseltamivir twice daily over 10 days. Participants in the Double dose arm received oseltamivir syrup at a dose ranging from 60 to 150 mg based on body weight, twice daily for children (1 to 12 years old) and oseltamivir capsules 150 mg twice daily for adolescents (>/=13 years old) over 10 days.
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
ng/mL
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 61.9
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 45.9
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 107
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 86.6

33. Secondary Outcome: Pharmacokinetics: Ctrough of Oseltamivir in Adolescents and Children
Description: Reported here are oseltamivir Ctrough data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: ng/mL
Groups:
- Adolescents and Children With Pharmacokinetic Evaluation: This analysis set comprises participants < 18 years from both arms in the study who underwent pharmacokinetic evaluation. Immunocompromised participants in the Conventional dose arm received oseltamivir syrup at doses ranging from 30 to 75 mg based on body weight, twice daily for children (1 to 12 years old) and oseltamivir capsules 75 mg twice daily for adolescents greater than or equal to (>/=) 13 years old or placebo-matched to oseltamivir twice daily over 10 days. Participants in the Double dose arm received oseltamivir syrup at a dose ranging from 60 to 150 mg based on body weight, twice daily for children (1 to 12 years old) and oseltamivir capsules 150 mg twice daily over 10 days.
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
ng/mL
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 2.84
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 3.37
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 6.65
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 3.88

34. Secondary Outcome: Pharmacokinetics: AUC0-12 at Steady State of Oseltamivir in Adolescents and Children
Description: AUC0-12 will be reported at steady state as ng*hr/mL. Reported here are oseltamivir AUC0-12 data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours on Day 6 or any day after the 11th dose
Population: The PKEP population comprised all subjects in the ITT population who had at least one valid post-dose drug concentration measurement at a scheduled visit time point.
Measure: Number; unit: ng*hr/mL
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
ng*hr/mL
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 229
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 171
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 425
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 339

35. Secondary Outcome: Pharmacokinetics: Tmax of Oseltamivir in Adolescents and Children
Description: Reported here are oseltamivir data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: hour
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
hour
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 1
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 1
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 1
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 1.25

36. Secondary Outcome: Pharmacokinetics: Cmax of Oseltamivir Carboxylate in Adolescents and Children
Description: Reported here are oseltamivir carboxylate Cmax data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: ng/mL
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
ng/mL
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 363
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 848
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 770
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 906

37. Secondary Outcome: Pharmacokinetics: Ctrough of Oseltamivir Carboxylate in Adolescents and Children
Description: Reported here are oseltamivir carboxylate Ctrough data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: ng/mL
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
ng/mL
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 215
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 459
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 445
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 464

38. Secondary Outcome: Pharmacokinetics: AUC0-12 at Steady State of Oseltamivir Carboxylate in Adolescents and Children
Description: AUC0-12 will be reported at steady state as ng*hr/mL. Reported here are oseltamivir carboxylate AUC0-12 data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: ng*hr/mL
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
ng*hr/mL
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 3550
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 8010
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 7460
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 8420

39. Secondary Outcome: Pharmacokinetics: Tmax of Oseltamivir Carboxylate in Adolescents and Children
Description: Reported here are oseltamivir carboxylate tmax data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: hour
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
hour
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 3.75
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 4
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 4
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 4

40. Secondary Outcome: Pharmacokinetics: Elimination Constant (ke) of Oseltamivir in Adolescents and Children
Description: Reported here are oseltamivir ke data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: 1/hr
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
1/hr
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 4.22
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 4.56
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 3.40
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 5.74

41. Secondary Outcome: Pharmacokinetics: Apparent Clearance (CL/F) of Oseltamivir in Adolescents and Children
Description: Reported here are oseltamivir CL/F data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: L/hr
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
L/hr
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 263
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 439
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 212
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 442

42. Secondary Outcome: Pharmacokinetics: Apparent Volume of Distribution (Vc/F) of Oseltamivir in Adolescents and Children
Description: Reported here are oseltamivir Vc/F data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: Liter (L)
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
Liter (L)
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 62.3
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 96.4
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 62.3
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 76.9

43. Secondary Outcome: Pharmacokinetics: Elimination Constant (ke) of Oseltamivir Carboxylate in Adolescents and Children
Description: Reported here are oseltamivir carboxylate ke data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: 1/hr
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
1/hr
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 2.01
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 1.12
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 1.44
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 2.12

44. Secondary Outcome: Pharmacokinetics: Apparent Clearance (CL/F), of Oseltamivir Carboxylate in Adolescents and Children
Description: Reported here are oseltamivir carboxylate CL/F data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: L/hr
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
L/hr
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 16.9
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 9.36
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 12.1
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 17.8

45. Secondary Outcome: Pharmacokinetics: Apparent Volume of Distribution (Vc/F) of Oseltamivir Carboxylate in Adolescents and Children
Description: Reported here are oseltamivir carboxylate Vc/F data for adolescents and children < 18 years. Individual data are provided as participants received different drug doses. Drug dose is indicated in the row title for each participant.
Time Frame: Pre-dose (30 minutes), 1.5, 4, 8 hours postdose on Day 6 or any day after the 11th dose
Population: as for outcome 19
Measure: Number; unit: Liter (L)
Arm/Group | Adolescents and Children With Pharmacokinetic Evaluation
Number analyzed (Participants) | 4
Liter (L)
  Conventional Dose: 60 mg: number analyzed (Participants) | 1
  Conventional Dose: 60 mg | 8.39
  Conventional Dose: 75 mg: number analyzed (Participants) | 1
  Conventional Dose: 75 mg | 8.39
  Double Dose: 90 mg: number analyzed (Participants) | 1
  Double Dose: 90 mg | 8.39
  Double Dose: 150 mg: number analyzed (Participants) | 1
  Double Dose: 150 mg | 8.39

ADVERSE EVENTS:
Time Frame: Baseline up to Day 40
Description: The safety population included all participants who received at least one treatment with study medication.
Arm/Group | Conventional Dose | Double Dose
All-Cause Mortality (participants affected / at risk) | 0/105 | 1/110
Serious Adverse Events (participants affected / at risk) | 8/105 | 10/110
Other Adverse Events (participants affected / at risk) | 23/105 | 35/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional Dose (N=105) | Double Dose (N=110)
Pneumonia (Infections and infestations) | 2 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional Dose (N=105) | Double Dose (N=110)
Diarrhoea (Gastrointestinal disorders) | 10 | 11
Nausea (Gastrointestinal disorders) | 10 | 14
Vomiting (Gastrointestinal disorders) | 10 | 12
Headache (Nervous system disorders) | 5 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2014-06-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT00545532/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT00545532/SAP_001.pdf